CLINICAL TRIAL: NCT06436079
Title: Evaluation of the Effectiveness of a Nursing Intervention Program in Reducing Anxiety in Users Who Perform Scheduled Sessions in the Hyperbaric Chamber
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Girona (Other)
Responsible Party: Principal Investigator, Lyudmila Andrusenko Kalchenko, Clinical professor, Universitat de Girona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 44519 ANSIETAT UMH
Record Dates: First submitted 2024-05-15; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Anxiety and Fear; Nurse's Role
Keywords: Anxiety; Nursing intervention; Hyperbaric chamber
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audiovisual educational program on treatment in a hyperbaric chamber (Experimental): The experimental group will receive a nursing educational intervention with an explanation, with audiovisual support, of the operation of the hyperbaric chamber.
  Interventions: Behavioral: Intervention group
- Usual intervention (Active Comparator): The control group will undergo the same procedure that is currently carried out, some basic explanations before entering the hyperbaric chamber.
  Interventions: Behavioral: Intervention group

INTERVENTIONS:
Behavioral: Intervention group — Patients who begin the first session in the hyperbaric chamber will receive a nursing educational intervention, with audiovisual support, about the operation of the chamber and aspects that must be taken into account once inside.

SUMMARY:
The objective of this experimental study is to determine if the application of a nursing educational intervention reduces the anxiety of patients who are going to undergo treatment in the hyperbaric chamber.

The researchers will compare the nursing educational intervention with the usual practice that is currently carried out in the unit for patients who are going to begin treatment in the hyperbaric chamber.

Participants will:

* Receive explanatory information through a camera triptych when the treatment is indicated.
* Come half an hour before the first session to receive a nursing educational intervention, with audiovisual support, on the operation of the camera.

DETAILED DESCRIPTION:
The objective of this experimental study is to determine if the application of a nursing educational intervention reduces the anxiety of patients who are going to undergo treatment in the hyperbaric chamber.

An educational intervention will be applied to the intervention group that will begin on the same day that the treatment is indicated. That day, you will be given an informative brochure about the most important aspects you should know about the hyperbaric chamber. On the first day of the session, you will be asked to come half an hour early to explain, in more detail, what the hyperbaric chamber consists of and important aspects that you should take into account.

The control group will receive the same intervention that is currently being carried out. Once treatment is prescribed in the chamber, they come on the first day and receive a brief explanation of how it works before entering.

ELIGIBILITY:
Inclusion Criteria:

* Results in the Pfeiffer questionnaire<2.
* That they understand Spanish or Catalan

Exclusion Criteria:

* That feel fear inside the hyperbaric chamber.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of anxiety measured with the STAI questionnaire. | First week of treatment in the hyperbaric chamber
  Feelings of fear, dread, and uneasiness that may occur as a reaction to stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Palamós, Palamós, Girona, Spain